CLINICAL TRIAL: NCT00393575
Title: Connect To Protect® Partnerships for Youth Prevention Interventions: Phase III
Brief Title: C2P Mobilization Intervention (Pilot)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); National Institute of Mental Health (NIMH) (NIH); National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: ATN 040
Record Dates: First submitted 2005-12-28; First posted 2006-10-30 (Estimated); Last update posted 2017-02-28 (Actual); Status verified 2016-07

CONDITIONS: HIV Infections
Keywords: HIV Prevention; HIV positive communities
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Community Mobilization (Experimental): The intervention population is defined as the community each site is attempting to mobilize.
  Interventions: Behavioral: Community Mobilization

INTERVENTIONS:
Behavioral: Community Mobilization — The intervention will consist of guiding C2P coalitions through a strategic planning process that will result in the development and implementation of a local action plan. The action plan will focus on changing structural elements of the affected communities that are believed to be associated with youth HIV acquisition and transmission. Each coalition's plan will include: (1) identification of potential community structural changes and specific steps for how to effect such changes; and (2) the selection of a community-level Centers for Disease Control and Prevention (CDC)-endorsed HIV prevention program.

SUMMARY:
Connect to Protect (C2P): Partnerships for Youth Prevention Interventions is a multi-site, three-phase project developed by the Adolescent Medicine Trials Network for HIV/AIDS Interventions (ATN). The overall goal of the project is to ultimately reduce HIV incidence and prevalence in youth 12-24 years old through a community mobilization intervention. This protocol (ATN 040) describes part one of Phase III. Part two of Phase III will be submitted as a separate protocol (ATN 041).

DETAILED DESCRIPTION:
The objective of Phase III is to initiate and complete a community mobilization intervention aimed at ultimately reducing HIV incidence and prevalence among youth. The intervention will consist of guiding C2P coalitions through a strategic planning process that will result in the development and implementation of a local action plan. The action plan will focus on changing structural elements of the affected communities that are believed to be associated with youth HIV acquisition and transmission. Each coalition's plan will include: (1) identification of potential community structural changes and specific steps for how to effect such changes; and (2) the selection of a community-level Centers for Disease Control and Prevention (CDC)-endorsed HIV prevention program. These activities will be described in this document. Details related to the training, technical assistance, adaptation, and implementation of the selected CDC program will be subsequently submitted for IRB review as part two of Phase III (ATN 041).

The intervention consists of community mobilization activities that are expected to lead to structural change and the adaptation and delivery of a CDC-endorsed HIV-prevention program. ATN/C2P staff at each site, with training and technical assistance from a C2P National Coordinating Center, will engage in a strategic planning process with their coalition members that results in the development and implementation of a local action plan.

The evaluation of the intervention will be within and across ATN/C2P sites implementing this protocol. For assessing the overall efficacy of the community mobilization intervention, data will be collected and analyzed from:

1. ATN/C2P site staff, in the form of systematic documentation of the community mobilization process and accomplishments (e.g., structural change achieved); and
2. Local public health departments and other similar sources of epidemiological information, as was done for generating Phase I epidemiologic profiles.

Duration: 4 years.

ELIGIBILITY:
Inclusion Criteria:

* Community each ATN/C2P site is attempting to mobilize

Exclusion Criteria:

* Non-ATN funded site

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2006-01; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Increasing levels of community mobilization will be associated with increasing levels of structural change over four years, as measured by new or modified programs, policies, and practices, within and across intervention communities. | Determined in analysis

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Ellen, MD, Study Chair — Johns Hopkins University Hospital
Locations (15):
- United States (14):
  - Children's Hospital of Los Angeles, Los Angeles, California
  - Univ of California at San Diego, San Diego, California
  - Univ of California at San Francisco, San Francisco, California
  - Children's Hosp. National Med. Ctr., Washington D.C., District of Columbia
  - Children's Diag. & Treatment Ctr., Fort Lauderdale, Florida
  - University of Miami, Miami, Florida
  - University of South Florida, Tampa, Florida
  - Stroger Hospital of Cook County, Chicago, Illinois
  - Tulane Medical Center, New Orleans, Louisiana
  - University of Maryland, Baltimore, Maryland
  - Childrens' Hospital Boston, Boston, Massachusetts
  - Mount Sinai Medical Center, New York, New York
  - Director, Adolescent AIDS Program, The Bronx, New York
  - The Children's Hosp. of Philadelphia, Philadelphia, Pennsylvania
- University Pediatric Hospital, San Juan, Puerto Rico

REFERENCES:
- See also: Website for the Adolescent Trials Network for HIV/AIDS Interventions — http://www.atnonline.org